CLINICAL TRIAL: NCT04298320
Title: Phase Ib/IIa Study of SHR-1210 Combined With AIN457 for Patients With Late Stage MSS CRC Who Failed Second-line and Above Treatment
Brief Title: A Trial of SHR-1210 in Combination With AIN457 in Patients With MSS CRC（SHR-1210-AIN457）
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqiao Zhang (Other)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, Director of the hospital, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNB001
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — camrelizumab; secukinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 + AIN457 (Experimental): SHR-1210 was administered 200mg iv every 2 weeks in combination with AIN457 150mg or 300mg ih every 2 weeks
  Interventions: Drug: SHR-1210; Drug: AIN 457

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 was administered 200mg iv every 2 weeks
Drug: AIN 457 — AIN457 was administered 150mg or 300mg ih every 2 weeks

SUMMARY:
This is a Phase Ib/IIa, Open-label, Investigator-initiated Trail of SHR-1210 (an Anti-PD-1 Inhibitor) in combination with AIN457 for patients with late stage MSS CRC who failed second-line and above treatment.

The main purpose of this study is to evaluate the safety, tolerability and RD of SHR-1210 combination with AIN457 as a treatment of MSS CRC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;

  1. Men or women aged 18-75 years;
  2. Patients with advanced colorectal cancer who failed to receive second-line or more standard treatment confirmed by pathology A)At least one measurable lesion that meets the RECIST v1.1 criteria; B)Microsatellite stability (MSS) required;
  3. ECOG score was 0 or 1;
  4. Have a life expectancy of at least 12 weeks;
  5. The functions of vital organs meet the following requirements:

     A) Sufficient bone marrow reserve: neutrophil absolute count ≥ 1.5x109/l, platelet ≥ 90x109 / L, hemoglobin ≥ 9 g / dl; B) Liver: plasma albumin ≥ 2.8g/dl; bilirubin ≤ 1.5 times of upper limit of normal value (ULN); ALT and AST ≤ 2.5uln, if there is liver metastasis, ALT and AST ≤ 5xuln; C) Kidney: serum creatinine ≤ 1.5 times ULN; D) Heart: left ventricular ejection fraction (LVEF) ≥ 50%; E) Coagulation: prothrombin time (PT) < 1.5 times ULN, INR ≤ 1.5 times ULN, APTT ≤ 1.5 times ULN; F) TSH ≤ ULN (if abnormal, FT3 and FT4 levels should be examined at the same time, if FT3 and FT4 levels are normal, they can be included in the group;
  6. Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 3 months after the last dose of study treatment;
  7. Patients can provide more than 8 pathological sections of previous and / or fresh tissue lesions;
  8. Volunteer to participate in this clinical trial, willing and able to follow the procedures related to clinical visit and research, understand the research procedures and have signed the informed consent.

Exclusion Criteria:

1. Those who have received anti-IL-17 or IL-23 drug treatment;
2. Have received PD-1 antibody treatment or other immunotherapy for PD-1/PD-L1;
3. Those who have received chemotherapy, molecular targeted drugs and anti-tumor drugs of traditional Chinese medicine within one month after the first use of the research drug;
4. The adverse reactions (except hair loss) caused by previous treatment did not recover to ≤ CTCAE level 1;
5. Those who have received radiotherapy and interventional treatment within one month after the first use of the study drug;
6. Those who have received major surgery or active ulcer or incomplete wound healing within one month after the first use of the study drug (excluding central vein catheterization, tumor tissue biopsy or nasogastric tube catheterization);
7. Those who received live attenuated vaccine within one month after the first use of the study drug or expected to receive live attenuated vaccine treatment during the study period;
8. Those who are expected to undergo elective surgery during the study period;
9. Those who received transfusion of blood products and injection of hematopoietic colony stimulating growth factor (such as G-CSF, GMCSF, M-CSF) within 14 days after the first use of the study drug;
10. Participants in another intervention clinical trial within one month after the first use of the study drug;
11. Within 5 years after the first use of the study drug or at the same time with other malignant tumors (except for cured skin basal cell carcinoma, cervical carcinoma in situ and ovarian cancer);
12. Patients with active autoimmune disease, or history of immunodeficiency and autoimmune disease, or disease history or syndrome requiring immunosuppressive drug treatment; (such as the following, but not limited to: asthma, idiopathic pulmonary fibrosis, bronchiolitis obliterans, colitis, drug pneumonia, idiopathic or interstitial pneumonia, autoimmune hepatitis, pituitary gland Inflammation, vasculitis, nephritis, uveitis, systemic lupus erythematosus, hyperthyroidism, hypothyroidism; patients with asthma in childhood have been completely relieved, and can be included in adults without any intervention, but asthma patients who need medical intervention with bronchodilator cannot be included);
13. Need systemic steroid hormone treatment;
14. Intestinal obstruction or fistula occurred within 3 months after the first use of the study drug;
15. Those who have ever had serious hypersensitivity reaction (defined as: the patients can't be relieved quickly after symptomatic treatment and / or infusion treatment; relapse after taking effect; leave the sequelae requiring hospitalization treatment); those who have allergic reaction to latex products;
16. People with tuberculosis (except old tuberculosis);
17. People infected with HBV or HCV or HIV;
18. There is active infection within 2 weeks after the first use of the study drug, or there is a history of persistent infection, chronic infection or recurrent infection, or there is active skin or soft tissue infection, including cellulitis, erysipelas, pustules, abscesses or fasciitis;
19. Patients with history of inflammatory bowel disease and / or active bowel disease;
20. People with uncontrollable pain;
21. It is known that there is metastasis of central nervous system or meninges;
22. Patients with uncontrollable pleural effusion, peritoneal effusion or pericardial effusion that need clinical intervention, such as those who need periodic repeated drainage or who have had serous effusion drainage recently (within 28 days before the first application);
23. Patients with uncontrollable chronic systemic diseases (such as severe chronic lung, liver, kidney or heart diseases); patients with arrhythmia, myocardial ischemia and long-term drug control; patients with acute myocardial infarction and current congestive heart failure in the previous year; patients with unstable angina or new angina within the last three months;
24. Hypertension patients whose systolic blood pressure is less than or equal to 160mhg and diastolic blood pressure is less than or equal to 100mhg;
25. Patients with known hereditary or acquired bleeding and thrombotic tendency (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism of spleen function, etc.); patients with bleeding tendency or undergoing thrombolysis or anticoagulation treatment; patients with significant clinical bleeding symptoms or clear bleeding tendency within 3 months before screening, such as daily cough/hemoptysis 2.5ml And above, gastrointestinal bleeding, esophageal and gastric varices with bleeding risk, and hemorrhagic gastric ulcer;
26. Those who have had the event of arteriovenous thrombosis within 6 months after the first use of the study drug, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc;
27. The subjects or their partners are or intend to be pregnant, and the subjects are or intend to breastfeed are not eligible for inclusion;
28. Those who have a clear history of neurological or mental disorders (such as depression); those whose objective conditions (including psychological state, family relationship, factors or geographical factors, etc.) make the subjects unable to complete the planned study or other factors that may lead to the forced termination of the study, and those who have combined treatment or laboratory examination abnormalities; 6 Who has a history of alcohol or drug abuse or has any uncontrolled medical condition within six months;
29. According to the judgment of the researchers, there are serious hazards to the safety of the subjects, or the accompanying diseases (such as severe diabetes) that affect the subjects to complete the study;
30. The researcher judged that other subjects did not conform to the enrollment of this experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
DLT (phase Ib) | Within four weeks after dosing
  Dose Limiting Toxicity
Incidence of Treatment-Emergent Adverse Events | from the first drug administration to within 90 days for the last SHR-1210 and AIN 457 dose
  adverse events/serious adverse events

SECONDARY OUTCOMES:
ORR | From the first drug administration up to two years
  Overall Response Rate
BOR | From the first drug administration up to two years
  Best Overall Response
DOR | From the first drug administration up to two years
  Duration of Response
DCR | From the first drug administration up to two years
  Disease Control Rate
PFS | From the first drug administration up to two years
  Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, PhD, Principal Investigator — Harbin Medical University Cancer Hosptital